CLINICAL TRIAL: NCT04952610
Title: An Open Label Extension Study of Etripamil Nasal Spray in Patients With Paroxysmal Supraventricular Tachycardia
Brief Title: Etripamil Nasal Spray in Patients With Paroxysmal Supraventricular Tachycardia
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Milestone Pharmaceuticals Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSP-2017-1278
Record Dates: First submitted 2021-04-23; First posted 2021-07-07 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-03

CONDITIONS: Paroxysmal Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: This is a multicenter study to enable patients with PVST to have continued access of etripamil NS. The study will only include patients who have participated in a Milestone Pharmaceuticals Inc. approved clinical research trial (NODE-301 Part 1, RAPID Study (NODE-301 Part 2), NODE-302, or NODE-303) of etripamil NS for PSVT. Patients who experienced any significant safety issues during participation in a previous study, as per Investigator's assessment, are excluded.
  This study is planned to continue until etripamil NS is commercially available for patients with PSVT or the study is terminated by the Sponsor for any reason.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etripamil NS 70 mg (Experimental): Self- administration of a dose of 70 mg of etripamil. Patients will be provided with a maximum of 4 pre-filled devices at a time. If the symptoms of PSVT persist 10 minutes after the first dose of etripamil NS 70 mg, a second dose of etripamil NS 70 mg can be self-administered by the patient. A second dose of etripamil NS 70 mg should be taken not earlier than 10, and not later than 15 minutes after the first dose.
  Interventions: Drug: Etripamil NS 70 mg; Device: Aptar Pharma Nasal Spray Bidose System

INTERVENTIONS:
Drug: Etripamil NS 70 mg — Etripamil will be administered via the Aptar Pharma Nasal Spray Bidose System.
Device: Aptar Pharma Nasal Spray Bidose System — Aptar Pharma Nasal Spray Bidose System will be supplied as prefilled devices packaged into child-resistant boxes with instructions for use provided in the study drug box.

SUMMARY:
This Open Label Extension study will enable eligible patients with Paroxysmal Supraventricular Tachycardia (PSVT) who have previously participated in a Milestone Pharmaceuticals clinical trial of etripamil NS for PSVT, to access continued treatment with etripamil NS, Patients who experienced any significant safety issues during participation period in a previous clinical trial of etripamil NS, as per Investigator's assessment , are excluded. This study will be conducted by Investigators who previously participated in a Milestone Pharmaceuticals clinical trial and are trained on the use of etripamil NS.

DETAILED DESCRIPTION:
Etripamil NS addresses an unmet medical need since there are currently no fast-acting products available for patient self-administered treatment of episodes of PSVT. The only currently available acute pharmacological therapy is IV treatment with adenosine or calcium channel blockers administered in a hospital or medically supervised environment. A self-administered product for PSVT would give patients the option to safely terminate acute episodes of PSVT without the need for a hospital visit and potential admission. An episodic treatment option may also allow selected patients to discontinue chronic prophylactic therapy with Class I, II (e.g., beta-blockers), III, and/or IV (e.g., calcium channel blockers) antiarrhythmic agents, thus avoiding the side effects and quality of life implications associated with these medications. Furthermore, patients weighing the risks of bridging therapy and an invasive catheter ablation procedure to address their PSVT would have the opportunity to consider episodic management with etripamil NS as a viable alternative treatment option.

The potential risks of study participation include those associated with exposure to etripamil NS. The side effect profile appears to be consistent with its expected pharmacology as a short-acting structural analog of verapamil, as well as with its delivery as moderately low pH nasal spray formulation. The most frequently reported (≥5% of subjects across all studies) AEs determined by the investigator to be possibly, probably, or definitely related to etripamil NS include headache, increased lacrimation, epistaxis, nasal congestion, nasal discomfort, rhinorrhea, sneezing and throat irritation.

Potential AEs, which have been rare or not observed in studies to date, include other cardiac arrhythmias, or AEs associated with drops in blood pressure (syncope, symptomatic hypotension).

The primary benefit of this study is that patients may be able to safely and rapidly terminate acute episodes of PSVT without the need for a hospital visit to receive IV medication. Patients may also be able to discontinue chronic prophylactic therapies they are taking for PSVT. Patients who are waiting for, ineligible, or unwilling to undergo ablation procedures may have an option for at-home treatment of their PSVT episodes.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for study participation if they meet all of the following criteria:

1. Has participated in a Milestone Pharmaceuticals Inc. clinical research trial of etripamil NS for the treatment of PSVT (NODE-301 Part1, RAPID (NODE-301 Part 2), NODE-302, or NODE-303.
2. Has signed the MSP-2017-1278 written informed consent;
3. Women of childbearing potential who are sexually active with a male partner who is not surgically sterile (i.e., vasectomy) must be willing to use at least 1 form of highly effective contraception from the time of signed informed consent until 7 days after the last administration of etripamil NS and must be willing to discontinue from the study should they become or plan to become pregnant.

   The following categories define females who are not considered to be of childbearing potential:
   * Postmenopausal females, defined as having amenorrhea for at least 12 months without an alternative medical cause; or
   * Premenopausal females with 1 of the following:

     1. Documented hysterectomy; or
     2. Documented bilateral salpingectomy; or
     3. Documented bilateral oophorectomy; or

   All females who do not meet at least one of the above criteria are considered to be of childbearing potential
4. Willing and able to comply with Investigator instructions on etripamil NS use and study requirements.

Exclusion Criteria:

A patient will be excluded from the study if they meet any of the following criteria:

1. History of allergic reaction to verapamil, etripamil, or any of the investigational medical components;
2. Current chronic therapy with digoxin, or any Class I or III antiarrhythmic drug. Patients may be eligible if these drugs are stopped at least five half-lives before enrollment. The only exception is oral amiodarone which must be stopped 30 days before enrollment;
3. History of ventricular pre-excitation, e.g., delta waves, Wolff-Parkinson-White syndrome;
4. History of a second- or third-degree atrioventricular block;
5. History of sick sinus syndrome and marked bradycardia (≤40 beats/minute);
6. History or evidence of severe ventricular arrhythmia (e.g. torsades de points, ventricular fibrillation, or sustained ventricular tachycardia)
7. Symptoms of congestive heart failure New York Heart Association Class II to IV;
8. Significant physical or psychiatric condition including alcoholism or drug abuse, which, in the opinion of the Investigator, could jeopardize the safety of the patient, or impede the patient's capacity to follow the study requirements;
9. Syncope due to an arrhythmic etiology or unexplained syncope during or after participation in an etripamil clinical research trial;
10. Is pregnant, breastfeeding, or is planning to become pregnant during the study;
11. History of acute coronary syndrome (without successful revascularization) or stroke within 6 months of enrollment;
12. Evidence of symptoms of hypotension within 24 hours following previous administration of etripamil, per Investigator's opinion.
13. Has experienced a significant safety issue related to study drug administration during participation in a previous etripamil study for PSVT, per the Investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The safety of self-administered etripamil Nasal Spray (NS) for treatment of episodes of PSVT outside of the clinical setting as assessed by patient-reported adverse events. | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (23):
- United States (17):
  - Site # 0160, Little Rock, Arkansas
  - Site # 1023, Vista, California
  - Site # 1083, West Hills, California
  - Site # 0102, Atlanta, Georgia
  - Site # 0137, Macon, Georgia
  - Site # 1115, Coeur d'Alene, Idaho
  - Site # 0149, Fort Wayne, Indiana
  - Site # 1025, West Des Moines, Iowa
  - Site # 1007, Salisbury, Maryland
  - Site # 0166, Lansing, Michigan
  - Site # 0114, New York, New York
  - Site # 1024, Canton, Ohio
  - Site # 0110, Toledo, Ohio
  - Site # 1123, Corvallis, Oregon
  - Site # 0105, Yardley, Pennsylvania
  - Site # 0122, Rapid City, South Dakota
  - Site # 1047, Austin, Texas
- Canada (6):
  - Site # 0213, Victoria, British Columbia
  - Site # 0210, Halifax, Nova Scotia
  - Site # 2006, Oshawa, Ontario
  - Site # 0204, Toronto, Ontario
  - Site # 0203, Montreal, Quebec
  - Site # 0205, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No